CLINICAL TRIAL: NCT02376790
Title: A Multicenter Double-Blind, Randomized Controlled Study of Etanercept and Methotrexate in Combination or as Monotherapy in Subjects With Psoriatic Arthritis
Brief Title: Etanercept and Methotrexate in Combination or as Monotherapy in Psoriatic Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20130207; 2014-004869-24 (EudraCT Number)
Record Dates: First submitted 2015-01-28; First posted 2015-03-03 (Estimated); Results first posted 2019-02-22 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis; Arthritis, Psoriasis; Etanercept; Enbrel; Methotrexate; Minimal Disease Activity
MeSH Terms: conditions — Arthritis, Psoriatic; Arthritis; Psoriasis | interventions — Etanercept; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Methotrexate Monotherapy (Active Comparator): Participants received oral methotrexate 20 mg weekly plus placebo to etanercept subcutaneous injection once a week for 48 weeks.
  Interventions: Drug: Methotrexate; Drug: Placebo to Etanercept
- Etanercept Monotherapy (Experimental): Participants received etanercept 50 mg weekly by subcutaneous injection plus oral placebo to methotrexate for 48 weeks.
  Interventions: Drug: Etanercept; Drug: Placebo to Methotrexate
- Methotrexate + Etanercept (Experimental): Participants received etanercept 50 mg a week by subcutaneous injection plus oral methotrexate 20 mg weekly for 48 weeks.
  Interventions: Drug: Etanercept; Drug: Methotrexate

INTERVENTIONS:
Drug: Etanercept — Etanercept was administered by subcutaneous injection once a week
  Other Names: Enbrel
  Arms: Etanercept Monotherapy; Methotrexate + Etanercept
Drug: Methotrexate — Methotrexate capsules taken orally once a week. Dosing was initiated at 10 mg weekly and titrated up to a final dose of 20 mg weekly over a 4-week period.
  Arms: Methotrexate + Etanercept; Methotrexate Monotherapy
Drug: Placebo to Etanercept — Placebo to etanercept was administered by subcutaneous injection once a week.
  Arms: Methotrexate Monotherapy
Drug: Placebo to Methotrexate — Placebo to methotrexate capsules taken orally once a week.
  Arms: Etanercept Monotherapy

SUMMARY:
The purpose of this study is to learn more about the role of etanercept alone or in combination with methotrexate on disease activity in adults with psoriatic arthritis.

DETAILED DESCRIPTION:
The study will consist of a 30-day screening period, a 48-week double-blind treatment period and a 30-day safety follow-up period.

At or after week 24, participants with an inadequate response could receive rescue therapy with etanercept plus methotrexate until the end of the treatment period.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject must have a diagnosis of psoriatic arthritis (PsA) by the Classification Criteria for Psoriatic Arthritis (CASPAR) criteria.
* Subject has ≥ 3 tender and ≥ 3 swollen joints at screening and at baseline.
* Subject has an active psoriatic skin lesion
* Subject is naïve to etanercept and any other biologic for the treatment for PsA or psoriasis.
* Subject has no prior use of methotrexate for PsA.
* Subject has no history of tuberculosis
* Subject has a negative test for tuberculosis, hepatitis B and C.

Exclusion Criteria:

* Subject has known history of alcoholic hepatitis, nonalcoholic steatohepatitis or immunodeficiency syndromes, including human immunodeficiency virus (HIV) infection.
* Subject has any active infection (including chronic or localized infections) for which anti-infectives were indicated within 4 weeks prior to the first dose of investigational product.
* Subject has a serious infection, defined as requiring hospitalization or intravenous anti-infectives within 8 weeks prior to the first dose of investigational product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 851 (Actual)
Dates: Start 2015-03-03 (Actual); Primary Completion 2018-01-09 (Actual); Study Completion 2018-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (125):
- United States (53):
  - Research Site, Tuscaloosa, Alabama
  - Research Site, Glendale, Arizona
  - Research Site, Mesa, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Escondido, California
  - Research Site, Hemet, California
  - Research Site, Los Angeles, California
  - Research Site, Mather, California
  - Research Site, Palm Desert, California
  - Research Site, San Francisco, California
  - Research Site, Santa Monica, California
  - Research Site, Thousand Oaks, California
  - Research Site, Tustin, California
  - Research Site, Aventura, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Kissimmee, Florida
  - Research Site, Ocoee, Florida
  - Research Site, Tampa, Florida
  - Research Site, Zephyrhills, Florida
  - Research Site, Meridian, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Springfield, Illinois
  - Research Site, Bowling Green, Kentucky
  - Research Site, Paducah, Kentucky
  - Research Site, Frederick, Maryland
  - Research Site, Hagerstown, Maryland
  - Research Site, Wheaton, Maryland
  - Research Site, Worcester, Massachusetts
  - Research Site, Lansing, Michigan
  - Research Site, Saint Clair Shores, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, Las Vegas, Nevada
  - Research Site, Lebanon, New Hampshire
  - Research Site, Clifton, New Jersey
  - Research Site, Freehold, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Wyomissing, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Dallas, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Chesapeake, Virginia
  - Research Site, Danville, Virginia
  - Research Site, Roanoke, Virginia
  - Research Site, Seattle, Washington
- Argentina (3):
  - Research Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Research Site, San Miguel de Tucumán, Tucumán Province
  - Research Site, Buenos Aires
- Bulgaria (5):
  - Research Site, Burgas
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sofia
- Canada (7):
  - Research Site, Surrey, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Québec, Quebec
  - Research Site, Trois-Rivières, Quebec
  - Research Site, Saskatoon, Saskatchewan
- Research Site, Santiago, Chile
- Czechia (6):
  - Research Site, Brno
  - Research Site, Ostrava-Trebovice
  - Research Site, Pardubice
  - Research Site, Prague
  - Research Site, Uherské Hradiště
  - Research Site, Zlín
- France (2):
  - Research Site, Lyon Cédex 3
  - Research Site, Poitiers
- Greece (2):
  - Research Site, Athens
  - Research Site, Thessaloniki
- Hungary (5):
  - Research Site, Budapest
  - Research Site, Nyíregyháza
  - Research Site, Szolnok
  - Research Site, Szombathely
  - Research Site, Veszprém
- Latvia (3):
  - Research Site, Liepāja
  - Research Site, Riga
  - Research Site, Valmiera
- Mexico (7):
  - Research Site, Mexicali, Baja California Norte
  - Research Site, Mexicalli, Baja California Norte
  - Research Site, Guadalajara, Jalisco
  - Research Site, Zapopan, Jalisco
  - Research Site, Monterrey, Nuevo León
  - Research Site, Culiacán, Sinaloa
  - Research Site, Chihuahua City
- Poland (4):
  - Research Site, Gdansk
  - Research Site, Lodz
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Portugal (2):
  - Research Site, Lisbon
  - Research Site, Ponte de Lima
- Puerto Rico (2):
  - Research Site, Ponce
  - Research Site, San Juan
- Russia (13):
  - Research Site, Chelyabinsk
  - Research Site, Kemerovo
  - Research Site, Kursk
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Orenburg
  - Research Site, Petrozavodsk
  - Research Site, Ryazan
  - Research Site, Saratov
  - Research Site, Smolensk
  - Research Site, Vladimir
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg
- South Africa (3):
  - Research Site, Panorama, Western Cape
  - Research Site, Pinelands, Western Cape
  - Research Site, Stellenbosch, Western Cape
- Spain (4):
  - Research Site, Córdoba, Andalusia
  - Research Site, Mérida, Extremadura
  - Research Site, A Coruña, Galicia
  - Research Site, Villajoyosa, Valencia
- United Kingdom (3):
  - Research Site, Bradford
  - Research Site, Dudley
  - Research Site, Nottingham

REFERENCES:
- [Background] Mease PJ, Gladman DD, Samad AS, Coates LC, Liu LXH, Aras GA, Collier DH, Chung JB. Design and rationale of the Study of Etanercept and Methotrexate in Combination or as Monotherapy in Subjects with Psoriatic Arthritis (SEAM-PsA). RMD Open. 2018 Feb 3;4(1):e000606. doi: 10.1136/rmdopen-2017-000606. eCollection 2018. PMID 29531787
- [Background] Mease PJ, Gladman DD, Collier DH, Ritchlin CT, Helliwell PS, Liu L, Kricorian G, Chung JB. Etanercept and Methotrexate as Monotherapy or in Combination for Psoriatic Arthritis: Primary Results From a Randomized, Controlled Phase III Trial. Arthritis Rheumatol. 2019 Jul;71(7):1112-1124. doi: 10.1002/art.40851. Epub 2019 May 28. PMID 30747501
- [Background] Strand V, Mease PJ, Maksabedian Hernandez EJ, Stolshek BS, Liu LXH, Collier DH, Kricorian G, Merola JF. Patient-reported outcomes data in patients with psoriatic arthritis from a randomised trial of etanercept and methotrexate as monotherapy or in combination. RMD Open. 2021 Jan;7(1):e001484. doi: 10.1136/rmdopen-2020-001484. PMID 33452180
- [Background] Coates LC, Merola JF, Mease PJ, Ogdie A, Gladman DD, Strand V, van Mens LJJ, Liu L, Yen PK, Collier DH, Kricorian G, Chung JB, Helliwell PS. Performance of composite measures used in a trial of etanercept and methotrexate as monotherapy or in combination in psoriatic arthritis. Rheumatology (Oxford). 2021 Mar 2;60(3):1137-1147. doi: 10.1093/rheumatology/keaa271. PMID 32864685
- [Background] Helliwell PS, Mease PJ, Kavanaugh A, Coates LC, Ogdie A, Deodhar A, Strand V, Kricorian G, Liu LXH, Collier D, Gladman DD. Impact of clinical domains other than arthritis on composite outcomes in psoriatic arthritis: comparison of treatment effects in the SEAM-PsA trial. RMD Open. 2022 Jul;8(2):e002366. doi: 10.1136/rmdopen-2022-002366. PMID 35863864
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 124 centers in Europe, Latin America, North America, and South Africa. Participants were enrolled from 03 March 2015 to 07 July 2017.
Pre-assignment Details: The study consisted of a 30-day screening period, a 48-week randomized double blind treatment period, and a 30-day safety follow-up period.
  Participants were randomly assigned in a 1:1:1 ratio to 1 of 3 treatment groups.
Groups:
- Etanercept + Methotrexate: Participants received etanercept 50 mg a week by subcutaneous injection and oral methotrexate 20 mg a week for 48 weeks.
Period: Overall Study
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Started | 284 | 284 | 283
Received Treatment | 282 | 284 | 282
Completed | 224 | 237 | 230
Not Completed | 60 | 47 | 53
Not completed — Withdrawal by Subject | 43 | 36 | 37
Not completed — Decision by Sponsor | 2 | 1 | 4
Not completed — Lost to Follow-up | 15 | 10 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate | Total
Number analyzed (Participants) | 284 | 284 | 283 | 851
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (13.1) | 48.5 (13.5) | 48.1 (12.7) | 48.4 (13.1)
Age, Customized [Count of Participants; unit: Participants]
  ≤ 65 years | 257 | 251 | 259 | 767
  > 65 years | 27 | 33 | 24 | 84
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 160 | 133 | 139 | 432
  Male | 124 | 151 | 144 | 419
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 58 | 70 | 69 | 197
  Not Hispanic or Latino | 226 | 214 | 214 | 654
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 | 11 | 8 | 30
  Asian | 3 | 1 | 1 | 5
  Black (or African American) | 4 | 0 | 3 | 7
  Mixed Race | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 2
  Other | 10 | 18 | 6 | 34
  White | 255 | 252 | 265 | 772
Body Mass Index (BMI) [Count of Participants; unit: Participants] — Population: Participants with available data
  Participants
    number analyzed (Participants) | 284 | 283 | 283 | 850
    ≤ 30 kg/m² | 146 | 153 | 160 | 459
    > 30 kg/m² | 138 | 130 | 123 | 391
Prior Use of Non-biologic Disease Modifying Antirheumatic Drugs (DMARDs) [Count of Participants; unit: Participants]
  Yes | 38 | 26 | 43 | 107
  No | 246 | 258 | 240 | 744
Duration of Psoriatic Arthritis Disease [Mean (Standard Deviation); unit: years] — Population: Participants with available data
  years
    number analyzed (Participants) | 231 | 222 | 231 | 684
    (all) | 3.64 (6.85) | 3.10 (5.96) | 2.96 (5.99) | 3.24 (6.28)
Swollen Joint Count [Mean (Standard Deviation); unit: joints] — A total of 66 joints were scored for presence or absence of swelling. Population: Participants with available data
  joints
    number analyzed (Participants) | 284 | 283 | 282 | 849
    (all) | 12.9 (9.9) | 11.5 (9.6) | 11.2 (9.1) | 11.9 (9.6)
Tender Joint Count [Mean (Standard Deviation); unit: joints] — A total of 68 joints were scored for presence or absence of tenderness. Population: Participants with available data
  joints
    number analyzed (Participants) | 284 | 283 | 282 | 849
    (all) | 20.9 (15.0) | 18.8 (14.5) | 20.0 (15.3) | 19.9 (14.9)
Physician Global Assessment of Disease Activity [Mean (Standard Deviation); unit: mm] — Assessed by the physician on a 100 mm visual analog scale (VAS), where 0 mm = No activity at all and 100 mm = Worst activity imaginable. Population: Participants with available data
  mm
    number analyzed (Participants) | 284 | 284 | 282 | 850
    (all) | 58.6 (19.4) | 58.3 (18.2) | 58.0 (17.8) | 58.3 (18.5)
Patient Global Assessment of Disease Activity [Mean (Standard Deviation); unit: mm] — Assessed by the participant on a 100 mm VAS, where 0 mm = No arthritis activity at all and 100 mm = Worst arthritis activity imaginable. Population: Participants with available data
  mm
    number analyzed (Participants) | 283 | 284 | 282 | 849
    (all) | 60.7 (22.5) | 62.9 (22.1) | 61.0 (20.8) | 61.5 (21.8)
Patient Global Assessment of Joint Pain [Mean (Standard Deviation); unit: mm] — Participants assessed their joint pain on a 100 mm VAS, where 0 mm = No pain at all and 100 mm = Worst pain imaginable. Population: Participants with available data
  mm
    number analyzed (Participants) | 283 | 284 | 282 | 849
    (all) | 56.1 (21.7) | 56.5 (22.3) | 55.7 (21.6) | 56.1 (21.8)
Disability Index of the Health Assessment Questionnaire (HAQ-DI) [Mean (Standard Deviation); unit: units on a scale] — The HAQ-DI is a patient-reported questionnaire consisting of 20 questions in eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and usual activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task are summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 283 | 284 | 282 | 849
    (all) | 1.3 (0.6) | 1.1 (0.6) | 1.2 (0.6) | 1.2 (0.6)
C-reactive Protein (CRP) Concentration [Mean (Standard Deviation); unit: mg/L] — C-reactive protein (CRP) is a protein found in blood. CRP levels rise in response to inflammation. Population: Participants with available data
  mg/L
    number analyzed (Participants) | 284 | 282 | 283 | 849
    (all) | 10.52 (16.29) | 10.72 (15.59) | 8.70 (11.65) | 9.98 (14.66)
Psoriatic Arthritis Disease Activity Score (PASDAS) [Median (Full Range); unit: units on a scale] — PASDAS is a measure of disease activity derived from the following:
  * Physician and patient global assessment of disease activity (0-100 VAS)
  * 68 tender joint count
  * 66 swollen joint count
  * Short Form-36 Questionnaire (SF-36) physical component summary (general health status on a scale from 0-100)
  * Tender dactylitis count (each digit assessed for tender dactylitis; total score 0-20)
  * Leeds enthesitis index (enthesitis assessed at 6 sites; total score of 0-6)
  * CRP
  The composite score is a weighted index where higher scores indicate more severe disease. Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 282 | 279 | 280 | 841
    (all) | 6.10 [2.2 to 9.1] | 6.02 [2.5 to 10.2] | 5.95 [3.0 to 9.4] | 6.02 [2.2 to 10.2]
Clinical Disease Activity Index (CDAI) [Mean (Standard Deviation); unit: units on a scale] — The Clinical Disease Activity Index (CDAI) is a composite index that is calculated as the sum of the following items:
  * 28 tender joint count,
  * 28 swollen joint count,
  * Patient's Global Assessment of Disease Activity measured on a 10 cm VAS, where 0 cm = lowest disease activity and 10 cm = highest;
  * Physician's Global Assessment of Disease Activity -measured on a 10 cm VAS, where 0 cm = lowest disease activity and 10 cm = highest.
  The CDAI score ranges from 0-76 where lower scores indicate less disease activity. Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 283 | 283 | 281 | 847
    (all) | 30.51 (13.26) | 28.45 (12.89) | 28.55 (12.71) | 29.17 (12.98)
Simplified Disease Activity Index (SDAI) [Mean (Standard Deviation); unit: units on a scale] — The Simplified Disease Activity Index (SDAI) is a composite index that is calculated as the sum of the following items:
  * 28 tender joint count,
  * 28 swollen joint count,
  * Patient's Global Assessment of Disease Activity measured on a 10 cm VAS, where 0 cm = lowest disease activity and 10 cm = highest;
  * Physician's Global Assessment of Disease Activity -measured on a 10 cm VAS, where 0 cm = lowest disease activity and 10 cm = highest.
  * CRP
  The SDAI score ranges from 0 to 86 with higher scores representing worse disease. Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 283 | 281 | 281 | 845
    (all) | 31.56 (13.52) | 29.52 (13.19) | 29.43 (12.90) | 30.17 (13.23)
Disease Activity Score 28 (DAS28) [Mean (Standard Deviation); unit: units on a scale] — The DAS28 measures the severity of disease at a specific time and is derived from the following variables:
  * 28 tender joint count
  * 28 swollen joint count
  * C-reactive protein (CRP) concentration
  * Patient's global assessment of disease activity, measured on a 100 mm VAS, where 0 mm = lowest disease activity and 100 mm = highest.
  DAS28(CRP) scores range from 0 to approximately 10, with the upper bound dependent on the highest possible level of CRP. Higher scores indicate higher disease activity. Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 283 | 281 | 281 | 845
    (all) | 4.93 (1.11) | 4.80 (1.13) | 4.75 (1.12) | 4.83 (1.12)
Medical Outcomes Health Survey Short Form 36 Items Version 2 (SF-36 v2) [Mean (Standard Deviation); unit: units on a scale] — The SF-36 is a health-related survey that assesses participant's quality of life and consists of 36 questions covering 8 health domains. Two summary component scores are calculated: mental component summary score (MCS) and physical component summary score (PCS). Each domain is scored by summing the individual items and transforming the scores into a 0 to 100 scale with higher scores indicating better health status or functioning. Population: Participants with available data
  units on a scale
    PCS: number analyzed (Participants) | 282 | 284 | 282 | 848
    PCS | 35.587 (8.411) | 37.835 (8.381) | 37.353 (9.243) | 36.927 (8.730)
    MCS: number analyzed (Participants) | 282 | 284 | 282 | 848
    MCS | 45.174 (12.073) | 45.107 (12.496) | 46.256 (11.236) | 45.511 (11.946)
Leeds Dactylitis Index (LDI) [Mean (Standard Deviation); unit: units on a scale] — The Leeds Dactylitis Index quantitatively measures dactylitis using the circumference of involved digits and control digits and tenderness of involved digits (on a scale from 0-3). The control digit is either the contralateral digit (digit on opposite hand or foot), or if the contralateral digit is also affected, from a standard reference table. The ratio of circumference between an affected digit and the control digit is multiplied by the tenderness score for the affected digit. The results from each involved digit are summed to provide the final LDI. A higher LDI indicates worse dactylitis. Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 284 | 283 | 282 | 849
    (all) | 56.89 (174.56) | 50.07 (137.20) | 44.11 (143.17) | 50.37 (152.47)
Spondyloarthritis Research Consortium of Canada (SPARCC) Enthesitis Index [Mean (Standard Deviation); unit: units on a scale] — The SPARCC enthesitis index assesses enthesitis at 18 sites for palpitation with a resultant total score of 0 to 16 (for scoring purposes, the inferior patella and tibial tuberosity are considered 1 site because of their anatomical proximity). Tenderness at each site is quantified on a dichotomous basis (0 = non-tender, 1 = tender). A higher count represents greater enthesitis burden. Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 284 | 283 | 282 | 849
    (all) | 3.9 (4.3) | 3.7 (4.3) | 4.1 (4.5) | 3.9 (4.4)
Percentage of Body Surface Area (BSA) Involved in Psoriasis [Mean (Standard Deviation); unit: percent body surface area] — The physician's assessment of the percentage of the participant's total body surface area involved with psoriasis. Population: Participants with available data
  percent body surface area | 12.68 (18.78) | 10.76 (14.66) | 10.74 (15.58) | 11.40 (16.44)
Static Physician Global Assessment (sPGA) [Mean (Standard Deviation); unit: units on a scale] — The static Physician Global Assessment of psoriasis (sPGA) evaluates the physician's global assessment of the participant's psoriasis based on severity of induration, scaling, and erythema. The sPGA is assessed on a scale from 0 to 5:
  0 = clear (no evidence of plaque elevation, erythema or scaling)
  1. = almost clear
  2. = mild
  3. = moderate
  4. = marked
  5. = severe Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 281 | 284 | 283 | 848
    (all) | 2.6 (1.1) | 2.6 (1.0) | 2.5 (1.0) | 2.6 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response at Week 24
Description: A positive ACR20 response is defined if the following 3 criteria for improvement from baseline were met:
  * ≥ 20% improvement in 68 tender joint count;
  * ≥ 20% improvement in 66 swollen joint count; and
  * ≥ 20% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of joint pain (measured on a 100 mm visual analog scale [VAS]);
    * Patient's global assessment of disease activity (measured on a 100 mm VAS);
    * Physician's global assessment of disease activity (measured on a 100 mm VAS);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]);
    * C-reactive protein concentration.
Time Frame: Baseline and week 24
Population: All randomized participants; missing postbaseline data were imputed using non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 284 | 284 | 283
percentage of participants | 50.7 | 60.9 | 65.0
Statistical Analysis 1: Comparison: Methotrexate Monotherapy vs Etanercept + Methotrexate; The primary hypothesis of this study is that etanercept plus methotrexate therapy and etanercept monotherapy are more efficacious than methotrexate monotherapy as measured by the percentage of participants with psoriatic arthritis achieving ACR 20 response at week 24; Test type: Superiority; p = 0.005, Cochran-Mantel-Haenszel — Adjusted p-value was obtained by applying a Bonferroni-based testing procedure for multiplicity adjustment to control the family-wise, two-sided type one error rate at 0.05; Cochran-Mantel-Haenszel test with baseline body mass index (≤ 30 kg/m² or > 30 kg/m²) and prior non-biologic DMARD treatment as stratification factors; Treatment Difference = 13.9, 95% CI 2-sided [5.8 to 22.0] — The risk difference was estimated using the Mantel-Haenszel estimate of common risk difference using the stratification factors described above
Statistical Analysis 2: Comparison: Methotrexate Monotherapy vs Etanercept Monotherapy; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.029, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Treatment Difference = 9.2, 95% CI 2-sided [1.0 to 17.3] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Percentage of Participants With a Minimal Disease Activity (MDA) Response at Week 24
Description: Minimal Disease Activity (MDA) is a measure of low disease activity specific for psoriatic arthritis (PsA) that incorporates measures of joint and entheseal inflammation, skin disease, patient reported outcomes and functional disability to assess disease activity. Participants were classified as achieving MDA if they fulfilled 5 of the following 7 outcome measures:
  * Tender joint count (0-68) ≤ 1
  * Swollen joint count (0-66) ≤ 1
  * Body surface area (BSA) involvement with psoriasis (0% to 100%) ≤ 3%
  * Patient global assessment of joint pain VAS (0-100) ≤ 15
  * Patient global assessment of disease activity VAS (0-100) ≤ 20
  * HAQ-DI (0-3) ≤ 0.5
  * Spondyloarthritis Research Consortium of Canada (SPARCC) enthesitis index (18 sites assessed for enthesitis with an overall score of 0 - 16) ≤ 1
Time Frame: Week 24
Population: All randomized participants; missing postbaseline data were imputed using non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 284 | 284 | 283
percentage of participants | 22.9 | 35.9 | 35.7
Statistical Analysis 1: Comparison: Methotrexate Monotherapy vs Etanercept + Methotrexate; The secondary hypothesis of this study was that etanercept plus methotrexate therapy and etanercept monotherapy are more efficacious than methotrexate monotherapy as measured by the percentage of participants with PsA achieving MDA response at week 24; Test type: Superiority; p = 0.005, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Treatment Difference = 12.2, 95% CI 2-sided [4.9 to 19.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Methotrexate Monotherapy vs Etanercept Monotherapy; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.005, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Treatment Difference = 11.6, 95% CI 2-sided [4.2 to 18.9] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response Over Time
Description: A positive ACR20 response is defined if the following 3 criteria for improvement from baseline were met:
  * ≥ 20% improvement in 68 tender joint count;
  * ≥ 20% improvement in 66 swollen joint count; and
  * ≥ 20% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of joint pain (measured on a 100 mm visual analog scale [VAS]);
    * Patient's global assessment of disease activity (measured on a 100 mm VAS);
    * Physician's global assessment of disease activity (measured on a 100 mm VAS);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]);
    * C-reactive protein.
Time Frame: Baseline and weeks 4, 8, 12, 16, 24, 36, and 48
Population: All randomized participants with non-missing data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 284 | 284 | 283
percentage of participants
  Week 4: number analyzed (Participants) | 280 | 280 | 276
  Week 4 | 25.0 | 44.3 | 46.4
  Week 8: number analyzed (Participants) | 271 | 274 | 268
  Week 8 | 46.5 | 60.2 | 60.8
  Week 12: number analyzed (Participants) | 267 | 267 | 263
  Week 12 | 46.8 | 65.5 | 70.3
  Week 16: number analyzed (Participants) | 253 | 256 | 248
  Week 16 | 58.5 | 69.5 | 71.8
  Week 24: number analyzed (Participants) | 253 | 256 | 256
  Week 24 | 56.9 | 67.6 | 71.9
  Week 36: number analyzed (Participants) | 243 | 248 | 240
  Week 36 | 66.3 | 77.0 | 74.2
  Week 48: number analyzed (Participants) | 229 | 237 | 230
  Week 48 | 70.7 | 83.1 | 80.4

4. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 50% (ACR50) Response Over Time
Description: A positive ACR50 response is defined if the following 3 criteria for improvement from baseline were met:
  * ≥ 50% improvement in 68 tender joint count;
  * ≥ 50% improvement in 66 swollen joint count; and
  * ≥ 50% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of joint pain (measured on a 100 mm visual analog scale [VAS]);
    * Patient's global assessment of disease activity (measured on a 100 mm VAS);
    * Physician's global assessment of disease activity (measured on a 100 mm VAS);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]);
    * C-reactive protein.
Time Frame: Baseline and weeks 4, 8, 12, 16, 24, 36, and 48
Population: All randomized participants with non-missing data at each time point
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 284 | 284 | 283
percentage of participants
  Week 4: number analyzed (Participants) | 281 | 279 | 276
  Week 4 | 6.0 | 16.5 | 18.8
  Week 8: number analyzed (Participants) | 272 | 275 | 269
  Week 8 | 15.1 | 31.3 | 30.1
  Week 12: number analyzed (Participants) | 267 | 267 | 263
  Week 12 | 16.9 | 40.4 | 39.2
  Week 16: number analyzed (Participants) | 253 | 256 | 251
  Week 16 | 29.2 | 43.8 | 43.4
  Week 24: number analyzed (Participants) | 252 | 257 | 256
  Week 24 | 30.6 | 44.4 | 45.7
  Week 36: number analyzed (Participants) | 244 | 246 | 241
  Week 36 | 41.8 | 57.3 | 56.0
  Week 48: number analyzed (Participants) | 229 | 238 | 231
  Week 48 | 49.3 | 63.0 | 60.2
Statistical Analysis 1: Comparison: Methotrexate Monotherapy vs Etanercept + Methotrexate; Analysis of the percentage of participants with an ACR50 response at week 24; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-value is unadjusted and considered descriptive; [statistical method as in outcome 1, analysis 1]; Treatment Difference = 14.7, 95% CI 2-sided [6.4 to 23.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Methotrexate Monotherapy vs Etanercept Monotherapy; Analysis of the percentage of participants with an ACR50 response at week 24; Test type: Superiority; p = 0.006, Cochran-Mantel-Haenszel — P-value is unadjusted and considered descriptive; [statistical method as in outcome 1, analysis 1]; Treatment Difference = 11.8, 95% CI 2-sided [3.4 to 20.2] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 70% (ACR70) Response Over Time
Description: A positive ACR70 response is defined if the following 3 criteria for improvement from baseline were met:
  * ≥ 70% improvement in 68 tender joint count;
  * ≥ 70% improvement in 66 swollen joint count; and
  * ≥ 70% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of joint pain (measured on a 100 mm visual analog scale [VAS]);
    * Patient's global assessment of disease activity (measured on a 100 mm VAS);
    * Physician's global assessment of disease activity (measured on a 100 mm VAS);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]);
    * C-reactive protein.
Time Frame: Baseline and weeks 4, 8, 12, 16, 24, 36, and 48
Population: All randomized participants with non-missing data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 284 | 284 | 283
percentage of participants
  Week 4: number analyzed (Participants) | 281 | 280 | 276
  Week 4 | 2.8 | 3.6 | 5.1
  Week 8: number analyzed (Participants) | 272 | 277 | 269
  Week 8 | 4.4 | 15.2 | 14.5
  Week 12: number analyzed (Participants) | 267 | 268 | 264
  Week 12 | 5.2 | 24.3 | 22.3
  Week 16: number analyzed (Participants) | 252 | 256 | 251
  Week 16 | 10.7 | 24.2 | 25.5
  Week 24: number analyzed (Participants) | 253 | 257 | 256
  Week 24 | 13.8 | 29.2 | 27.7
  Week 36: number analyzed (Participants) | 245 | 247 | 242
  Week 36 | 19.6 | 38.5 | 33.5
  Week 48: number analyzed (Participants) | 230 | 237 | 232
  Week 48 | 25.2 | 39.7 | 39.7
Statistical Analysis 1: Comparison: Methotrexate Monotherapy vs Etanercept + Methotrexate; Analysis of the percentage of participants with an ACR70 response at week 24; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-value is unadjusted and considered descriptive; [statistical method as in outcome 1, analysis 1]; Treatment Difference = 13.4, 95% CI 2-sided [6.5 to 20.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Methotrexate Monotherapy vs Etanercept Monotherapy; Analysis of the percentage of participants with an ACR70 response at week 24; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-value is unadjusted and considered descriptive; [statistical method as in outcome 1, analysis 1]; Treatment Difference = 13.7, 95% CI 2-sided [6.7 to 20.7] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Change From Baseline in Tender Joint Count Over Time
Description: The tender joint count is an assessment of the pain and/or tenderness of 68 joints using a 0 to 1 point scale (0 = none, 1 = present). The total tender joint count is calculated by summing the number of joints with present tenderness.
Time Frame: Baseline and weeks 4, 8, 12, 16, 24, 36, and 48
Population: All randomized participants with non-missing data at each time point
Measure: Mean (Standard Error); unit: tender joints
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 284 | 284 | 283
tender joints
  Week 4: number analyzed (Participants) | 280 | 279 | 277
  Week 4 | -5.7 (0.6) | -6.4 (0.6) | -7.4 (0.6)
  Week 8: number analyzed (Participants) | 271 | 276 | 269
  Week 8 | -7.8 (0.7) | -8.9 (0.6) | -9.4 (0.7)
  Week 12: number analyzed (Participants) | 266 | 267 | 264
  Week 12 | -9.7 (0.7) | -9.8 (0.7) | -10.8 (0.7)
  Week 16: number analyzed (Participants) | 253 | 257 | 251
  Week 16 | -10.0 (0.7) | -10.9 (0.7) | -11.9 (0.8)
  Week 24: number analyzed (Participants) | 253 | 257 | 257
  Week 24 | -10.8 (0.8) | -10.9 (0.8) | -11.0 (0.9)
  Week 36: number analyzed (Participants) | 245 | 248 | 243
  Week 36 | -13.5 (0.8) | -12.7 (0.8) | -12.9 (0.9)
  Week 48: number analyzed (Participants) | 230 | 239 | 232
  Week 48 | -14.5 (0.8) | -13.9 (0.8) | -12.9 (0.9)

7. Secondary Outcome: Change From Baseline in Swollen Joint Count Over Time
Description: The swollen joint count is an assessment of the swelling of 66 joints using a 0 to 1 point scale (0 = none, 1 = present). The total swollen joint count is calculated by summing the number of joints with present swelling.
Time Frame: Baseline and weeks 4, 8, 12, 16, 24, 36, and 48
Population: All randomized participants with non-missing data at each time point
Measure: Mean (Standard Error); unit: swollen joints
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 284 | 284 | 283
swollen joints
  Week 4: number analyzed (Participants) | 280 | 279 | 277
  Week 4 | -4.1 (0.4) | -4.8 (0.3) | -4.7 (0.4)
  Week 8: number analyzed (Participants) | 271 | 276 | 269
  Week 8 | -5.4 (0.5) | -6.2 (0.4) | -6.5 (0.4)
  Week 12: number analyzed (Participants) | 266 | 267 | 264
  Week 12 | -6.6 (0.5) | -6.8 (0.4) | -7.2 (0.4)
  Week 16: number analyzed (Participants) | 253 | 257 | 251
  Week 16 | -7.0 (0.5) | -7.3 (0.4) | -7.8 (0.4)
  Week 24: number analyzed (Participants) | 253 | 257 | 257
  Week 24 | -7.0 (0.5) | -7.6 (0.5) | -7.7 (0.5)
  Week 36: number analyzed (Participants) | 245 | 248 | 243
  Week 36 | -9.2 (0.5) | -9.0 (0.5) | -8.4 (0.5)
  Week 48: number analyzed (Participants) | 230 | 239 | 232
  Week 48 | -9.6 (0.5) | -9.2 (0.5) | -8.7 (0.5)

8. Secondary Outcome: Change From Baseline in Physician Global Assessment of Disease Activity Over Time
Description: A global assessment of the participant's arthritis assessed by the physician on a 100 mm visual analog scale (VAS) where 0 mm = No activity at all and 100 mm = Worst activity imaginable.
Time Frame: Baseline and weeks 4, 8, 12, 16, 24, 36, and 48
Population: All randomized participants with non-missing data at each time point
Measure: Mean (Standard Error); unit: mm
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 284 | 284 | 283
mm
  Week 4: number analyzed (Participants) | 278 | 278 | 277
  Week 4 | -16.8 (1.2) | -23.1 (1.2) | -22.8 (1.3)
  Week 8: number analyzed (Participants) | 271 | 277 | 269
  Week 8 | -25.0 (1.4) | -29.7 (1.4) | -30.4 (1.4)
  Week 12: number analyzed (Participants) | 266 | 267 | 264
  Week 12 | -26.8 (1.6) | -32.7 (1.6) | -33.9 (1.3)
  Week 16: number analyzed (Participants) | 251 | 257 | 252
  Week 16 | -30.3 (1.7) | -34.9 (1.5) | -36.2 (1.4)
  Week 24: number analyzed (Participants) | 250 | 257 | 257
  Week 24 | -29.6 (1.8) | -35.7 (1.7) | -35.8 (1.6)
  Week 36: number analyzed (Participants) | 241 | 246 | 241
  Week 36 | -37.1 (1.7) | -42.8 (1.5) | -39.9 (1.5)
  Week 48: number analyzed (Participants) | 229 | 239 | 232
  Week 48 | -41.4 (1.5) | -43.8 (1.4) | -41.5 (1.6)

9. Secondary Outcome: Change From Baseline in Patient Global Assessment of Disease Activity Over Time
Description: A global assessment of the participant's arthritis, assessed by the participant on a 100 mm VAS where 0 mm = No arthritis activity at all and 100 mm = Worst arthritis activity imaginable.
Time Frame: Baseline and weeks 4, 8, 12, 16, 24, 36, and 48
Population: All randomized participants with non-missing data at each time point
Measure: Mean (Standard Error); unit: mm
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 284 | 284 | 283
mm
  Week 4: number analyzed (Participants) | 280 | 281 | 277
  Week 4 | -11.0 (1.5) | -21.9 (1.6) | -21.0 (1.5)
  Week 8: number analyzed (Participants) | 271 | 277 | 269
  Week 8 | -15.6 (1.6) | -27.3 (1.6) | -26.4 (1.6)
  Week 12: number analyzed (Participants) | 266 | 268 | 264
  Week 12 | -18.6 (1.6) | -29.9 (1.7) | -28.0 (1.7)
  Week 16: number analyzed (Participants) | 252 | 257 | 250
  Week 16 | -22.7 (1.7) | -30.9 (1.7) | -29.3 (1.7)
  Week 24: number analyzed (Participants) | 252 | 258 | 257
  Week 24 | -23.0 (1.8) | -32.3 (1.7) | -29.6 (1.8)
  Week 36: number analyzed (Participants) | 243 | 248 | 241
  Week 36 | -26.0 (1.8) | -36.4 (1.8) | -32.4 (1.8)
  Week 48: number analyzed (Participants) | 228 | 238 | 232
  Week 48 | -28.9 (1.9) | -38.8 (1.7) | -33.3 (1.9)

10. Secondary Outcome: Change From Baseline in Patient Global Assessment of Joint Pain Over Time
Description: A global assessment of the severity of the participant's joint pain, assessed by the participant on a 100 mm VAS where 0 mm = No pain at all and 100 mm = Worst pain imaginable.
Time Frame: Baseline and weeks 4, 8, 12, 16, 24, 36, and 48
Population: All randomized participants with non-missing data at each time point
Measure: Mean (Standard Error); unit: mm
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 284 | 284 | 283
mm
  Week 4: number analyzed (Participants) | 280 | 281 | 277
  Week 4 | -8.9 (1.4) | -18.4 (1.5) | -18.5 (1.6)
  Week 8: number analyzed (Participants) | 271 | 277 | 269
  Week 8 | -14.5 (1.5) | -23.5 (1.5) | -24.0 (1.5)
  Week 12: number analyzed (Participants) | 266 | 268 | 264
  Week 12 | -16.0 (1.6) | -24.1 (1.7) | -24.9 (1.6)
  Week 16: number analyzed (Participants) | 252 | 257 | 250
  Week 16 | -20.9 (1.7) | -25.9 (1.7) | -25.6 (1.7)
  Week 24: number analyzed (Participants) | 252 | 258 | 257
  Week 24 | -20.6 (1.7) | -26.4 (1.7) | -26.9 (1.7)
  Week 36: number analyzed (Participants) | 243 | 248 | 241
  Week 36 | -23.9 (1.7) | -31.5 (1.7) | -28.8 (1.8)
  Week 48: number analyzed (Participants) | 228 | 238 | 232
  Week 48 | -27.2 (1.8) | -32.5 (1.7) | -31.1 (1.8)

11. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire- Disability Index (HAQ-DI) Over Time
Description: The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire consisting of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and usual activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task are summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. Negative mean changes from Baseline in the overall score indicate improvement in functional ability.
Time Frame: Baseline and weeks 4, 8, 12, 16, 24, 36, and 48
Population: All randomized participants with non-missing data at each time point
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 284 | 284 | 283
units on a scale
  Week 4: number analyzed (Participants) | 280 | 281 | 277
  Week 4 | -0.188 (0.024) | -0.266 (0.024) | -0.306 (0.029)
  Week 8: number analyzed (Participants) | 271 | 276 | 269
  Week 8 | -0.277 (0.029) | -0.365 (0.031) | -0.403 (0.032)
  Week 12: number analyzed (Participants) | 266 | 268 | 264
  Week 12 | -0.310 (0.030) | -0.404 (0.029) | -0.450 (0.033)
  Week 16: number analyzed (Participants) | 252 | 257 | 250
  Week 16 | -0.378 (0.036) | -0.454 (0.033) | -0.483 (0.036)
  Week 24: number analyzed (Participants) | 252 | 258 | 257
  Week 24 | -0.412 (0.036) | -0.444 (0.035) | -0.468 (0.038)
  Week 36: number analyzed (Participants) | 243 | 248 | 241
  Week 36 | -0.452 (0.038) | -0.496 (0.039) | -0.548 (0.040)
  Week 48: number analyzed (Participants) | 228 | 238 | 232
  Week 48 | -0.526 (0.041) | -0.557 (0.038) | -0.554 (0.041)

12. Secondary Outcome: Change From Baseline in C-reactive Protein Concentration Over Time
Description: C-reactive protein (CRP) is a specific measure of inflammatory activity.
Time Frame: Baseline and weeks 4, 8, 12, 16, 24, 36, and 48
Population: All randomized participants with non-missing data at each time point
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 284 | 284 | 283
mg/L
  Week 4: number analyzed (Participants) | 275 | 265 | 256
  Week 4 | -0.93 (0.93) | -5.91 (1.01) | -5.49 (0.74)
  Week 8: number analyzed (Participants) | 270 | 265 | 257
  Week 8 | -2.31 (0.90) | -7.51 (0.94) | -5.19 (0.88)
  Week 12: number analyzed (Participants) | 262 | 255 | 247
  Week 12 | -3.36 (0.84) | -7.38 (0.99) | -5.71 (0.82)
  Week 16: number analyzed (Participants) | 248 | 246 | 241
  Week 16 | -2.81 (0.82) | -7.40 (1.03) | -5.59 (0.85)
  Week 24: number analyzed (Participants) | 246 | 249 | 247
  Week 24 | -2.60 (0.91) | -6.91 (1.15) | -5.82 (0.70)
  Week 36: number analyzed (Participants) | 236 | 234 | 230
  Week 36 | -4.16 (0.96) | -7.36 (1.13) | -5.82 (0.80)
  Week 48: number analyzed (Participants) | 223 | 226 | 219
  Week 48 | -4.88 (1.03) | -7.45 (1.10) | -5.81 (0.95)

13. Secondary Outcome: Percentage of Participants With a American Minimal Disease Activity (MDA) Response Over Time
Description: as for outcome 2
Time Frame: Weeks 4, 8, 12, 24, 36, and 48
Population: All randomized participants with non-missing data at each time point
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 284 | 284 | 283
percentage of participants
  Week 4: number analyzed (Participants) | 281 | 280 | 278
  Week 4 | 5.7 | 11.1 | 12.6
  Week 8: number analyzed (Participants) | 271 | 276 | 270
  Week 8 | 3.0 | 9.4 | 7.4
  Week 12: number analyzed (Participants) | 267 | 268 | 265
  Week 12 | 11.6 | 29.9 | 29.1
  Week 24: number analyzed (Participants) | 253 | 258 | 258
  Week 24 | 25.7 | 39.5 | 39.1
  Week 36: number analyzed (Participants) | 244 | 248 | 242
  Week 36 | 30.3 | 43.5 | 46.7
  Week 48: number analyzed (Participants) | 229 | 238 | 233
  Week 48 | 35.8 | 51.3 | 53.2

14. Secondary Outcome: Change From Baseline in Psoriatic Arthritis Disease Activity Score (PASDAS) Over Time
Description: PASDAS is a measure of disease activity derived from the following variables:
  * Physician and patient global assessment of disease activity (assessed on a 0-100 VAS)
  * 68 tender joint count
  * 66 swollen joint count
  * Short Form-36 Questionnaire (SF-36) physical component summary (general health status on a scale from 0-100)
  * Tender dactylitis count (each digit assessed for tender dactylitis; total score 0-20)
  * Leeds enthesitis index (enthesitis assessed at 6 sites; total score of 0-6)
  * CRP level (mg/L)
  The composite score is a weighted index where higher scores indicate more severe disease.
Time Frame: Baseline and weeks 12, 24, 36, and 48
Population: All randomized participants with non-missing data at each time point
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 284 | 284 | 283
units on a scale
  Week 12: number analyzed (Participants) | 261 | 263 | 261
  Week 12 | -1.63 (0.08) | -2.32 (0.09) | -2.37 (0.09)
  Week 24: number analyzed (Participants) | 246 | 250 | 255
  Week 24 | -1.98 (0.10) | -2.64 (0.10) | -2.63 (0.11)
  Week 36: number analyzed (Participants) | 234 | 238 | 232
  Week 36 | -2.46 (0.10) | -3.10 (0.10) | -2.95 (0.11)
  Week 48: number analyzed (Participants) | 226 | 232 | 229
  Week 48 | -2.70 (0.10) | -3.23 (0.09) | -3.10 (0.11)
Statistical Analysis 1: Comparison: Methotrexate Monotherapy vs Etanercept + Methotrexate; Analysis of change from baseline in PASDAS at week 24; Test type: Superiority; p < 0.001, ANCOVA — P-value is unadjusted and considered descriptive; ANCOVA model adjusted for baseline BMI status (≤ 30 kg/m² or > 30 kg/m²) and prior non-biologic DMARD use; LS Mean Treatment Difference = -0.62, 95% CI 2-sided [-0.91 to -0.34], Standard Error of Mean 0.14 — Methotrexate Monotherapy is the reference
Statistical Analysis 2: Comparison: Methotrexate Monotherapy vs Etanercept Monotherapy; Analysis of change from baseline in PASDAS at week 24; Test type: Superiority; p < 0.001, ANCOVA — P-value is unadjusted and considered descriptive; ANCOVA model adjusted for baseline BMI status (≤ 30 kg/m² or >30 kg/m²) and prior non-biologic DMARD use; LS Mean Treatment Difference = -0.63, 95% CI 2-sided [-0.92 to -0.34], Standard Error of Mean 0.15 — Methotrexate Monotherapy is the reference

15. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) Over Time
Description: The Clinical Disease Activity Index (CDAI) is a composite index that is calculated as the sum of the following items:
  * 28 tender joint count,
  * 28 swollen joint count,
  * Patient's Global Assessment of Disease Activity measured on a 10 cm VAS, where 0 cm = lowest disease activity and 10 cm = highest;
  * Physician's Global Assessment of Disease Activity -measured on a 10 cm VAS, where 0 cm = lowest disease activity and 10 cm = highest.
  The CDAI score ranges from 0-76 where lower scores indicate less disease activity.
Time Frame: Baseline and weeks 4, 8, 12, 16, 24, 36, and 48
Population: All randomized participants with non-missing data at each time point
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 284 | 284 | 283
units on a scale
  Week 4: number analyzed (Participants) | 276 | 277 | 276
  Week 4 | -8.38 (0.62) | -10.59 (0.61) | -10.68 (0.60)
  Week 8: number analyzed (Participants) | 270 | 276 | 268
  Week 8 | -11.56 (0.73) | -14.13 (0.66) | -14.56 (0.65)
  Week 12: number analyzed (Participants) | 265 | 266 | 263
  Week 12 | -13.93 (0.74) | -15.61 (0.75) | -16.12 (0.71)
  Week 16: number analyzed (Participants) | 250 | 256 | 248
  Week 16 | -15.20 (0.80) | -16.49 (0.70) | -17.37 (0.76)
  Week 24: number analyzed (Participants) | 249 | 257 | 256
  Week 24 | -15.74 (0.85) | -17.12 (0.78) | -16.43 (0.85)
  Week 36: number analyzed (Participants) | 240 | 246 | 239
  Week 36 | -18.90 (0.76) | -19.79 (0.76) | -18.86 (0.79)
  Week 48: number analyzed (Participants) | 228 | 238 | 231
  Week 48 | -20.16 (0.80) | -20.78 (0.75) | -19.35 (0.83)
Statistical Analysis 1: Comparison: Methotrexate Monotherapy vs Etanercept + Methotrexate; Analysis of change from baseline in CDAI at week 24; Test type: Superiority; p = 0.59, ANCOVA — P-value is unadjusted and considered descriptive; ANCOVA model adjusted for baseline BMI status (≤ 30 kg/m² or > 30 kg/m²) and prior non-biologic DMARD use; LS Mean Treatment Difference = -0.63, 95% CI 2-sided [-2.93 to 1.68], Standard Error of Mean 1.18 — Methotrexate Monotherapy is the reference
Statistical Analysis 2: Comparison: Methotrexate Monotherapy vs Etanercept Monotherapy; Analysis of change from baseline in CDAI at week 24; Test type: Superiority; p = 0.26, ANCOVA — P-value is unadjusted and considered descriptive; ANCOVA model adjusted for baseline BMI status (≤ 30 kg/m² or > 30 kg/m²) and prior non-biologic DMARD use; LS Mean Treatment Difference = -1.32, 95% CI 2-sided [-3.63 to 0.99], Standard Error of Mean 1.18 — Methotrexate Monotherapy is the reference

16. Secondary Outcome: Change From Baseline in Simplified Disease Activity Index (SDAI) Over Time
Description: The Simplified Disease Activity Index (SDAI) is a composite index that is calculated as the sum of the following items:
  * 28 tender joint count,
  * 28 swollen joint count,
  * Patient's Global Assessment of Disease Activity measured on a 10 cm VAS, where 0 cm = lowest disease activity and 10 cm = highest;
  * Physician's Global Assessment of Disease Activity -measured on a 10 cm VAS, where 0 cm = lowest disease activity and 10 cm = highest.
  * CRP
  The SDAI score ranges from 0 to 86 with higher scores representing worse disease.
Time Frame: Baseline and weeks 4, 8, 12, 16, 24, 36, and 48
Population: All randomized participants with non-missing data at each time point
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 284 | 284 | 283
units on a scale
  Week 4: number analyzed (Participants) | 275 | 273 | 273
  Week 4 | -8.38 (0.62) | -11.12 (0.62) | -11.18 (0.61)
  Week 8: number analyzed (Participants) | 270 | 272 | 267
  Week 8 | -11.77 (0.72) | -14.92 (0.69) | -15.14 (0.66)
  Week 12: number analyzed (Participants) | 264 | 264 | 263
  Week 12 | -14.32 (0.75) | -16.44 (0.77) | -16.67 (0.73)
  Week 16: number analyzed (Participants) | 248 | 253 | 246
  Week 16 | -15.55 (0.81) | -17.25 (0.72) | -17.79 (0.78)
  Week 24: number analyzed (Participants) | 248 | 253 | 256
  Week 24 | -15.96 (0.86) | -17.75 (0.81) | -17.01 (0.87)
  Week 36: number analyzed (Participants) | 239 | 242 | 235
  Week 36 | -19.27 (0.77) | -20.50 (0.78) | -19.46 (0.82)
  Week 48: number analyzed (Participants) | 228 | 234 | 229
  Week 48 | -20.65 (0.81) | -21.61 (0.77) | -19.94 (0.87)
Statistical Analysis 1: Comparison: Methotrexate Monotherapy vs Etanercept + Methotrexate; Analysis of change from baseline in SDAI at week 24; Test type: Superiority; p = 0.41, ANCOVA — P-value is unadjusted and considered descriptive; ANCOVA model adjusted for baseline BMI status (≤ 30 kg/m² or > 30 kg/m²) and prior non-biologic DMARD use; LS Mean Treatment Difference = -0.98, 95% CI 2-sided [-3.35 to 1.38], Standard Error of Mean 1.20 — Methotrexate Monotherapy is the reference
Statistical Analysis 2: Comparison: Methotrexate Monotherapy vs Etanercept Monotherapy; Analysis of change from baseline in SDAI at week 24; Test type: Superiority; p = 0.15, ANCOVA — P-value is unadjusted and considered descriptive; ANCOVA model adjusted for baseline BMI status (≤ 30 kg/m² or > 30 kg/m²) and prior non-biologic DMARD use; LS Mean Treatment Difference = -1.72, 95% CI 2-sided [-4.09 to 0.65], Standard Error of Mean 1.21 — Methotrexate Monotherapy is the reference

17. Secondary Outcome: Change From Baseline in the Disease Activity Score 28 (DAS28) Over Time
Description: The DAS28 measures the severity of disease at a specific time and is derived from the following variables:
  * 28 tender joint count
  * 28 swollen joint count
  * C-reactive protein (CRP)
  * Patient's global assessment of disease activity, measured on a 100 mm VAS, where 0 mm = lowest disease activity and 100 mm = highest.
  DAS28(CRP) scores range from 0 to approximately 10, with the upper bound dependent on the highest possible level of CRP. A DAS28 score higher than 5.1 indicates high disease activity, a DAS28 score less than 3.2 indicates low disease activity, and a DAS28 score less than 2.6 indicates clinical remission.
Time Frame: Baseline and weeks 4, 8, 12, 16, 24, 36, and 48
Population: All randomized participants with non-missing data at each time point
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 284 | 284 | 283
units on a scale
  Week 4: number analyzed (Participants) | 278 | 275 | 273
  Week 4 | -0.73 (0.05) | -1.18 (0.06) | -1.21 (0.06)
  Week 8: number analyzed (Participants) | 270 | 272 | 267
  Week 8 | -1.05 (0.06) | -1.64 (0.07) | -1.61 (0.07)
  Week 12: number analyzed (Participants) | 264 | 265 | 263
  Week 12 | -1.34 (0.06) | -1.78 (0.08) | -1.80 (0.08)
  Week 16: number analyzed (Participants) | 250 | 253 | 246
  Week 16 | -1.47 (0.07) | -1.90 (0.08) | -1.92 (0.08)
  Week 24: number analyzed (Participants) | 251 | 253 | 256
  Week 24 | -1.55 (0.08) | -1.97 (0.08) | -1.86 (0.08)
  Week 36: number analyzed (Participants) | 242 | 244 | 236
  Week 36 | -1.88 (0.07) | -2.25 (0.08) | -2.20 (0.09)
  Week 48: number analyzed (Participants) | 228 | 234 | 229
  Week 48 | -2.04 (0.07) | -2.38 (0.08) | -2.23 (0.09)
Statistical Analysis 1: Comparison: Methotrexate Monotherapy vs Etanercept + Methotrexate; Analysis of change from baseline in DAS28 at week 24; Test type: Superiority; p = 0.010, ANCOVA — P-value is unadjusted and considered descriptive; ANCOVA model adjusted for baseline BMI status (≤ 30 kg/m² or >30 kg/m²) and prior non-biologic DMARD use; LS Mean Treatment Difference = -0.29, 95% CI 2-sided [-0.52 to -0.07], Standard Error of Mean 0.11 — Methotrexate Monotherapy is the reference
Statistical Analysis 2: Comparison: Methotrexate Monotherapy vs Etanercept Monotherapy; Analysis of change from baseline in DAS28 at week 24; Test type: Superiority; p < 0.001, ANCOVA — P-value is unadjusted and considered descriptive; ANCOVA model adjusted for baseline BMI status (≤ 30 kg/m² or >30 kg/m²) and prior non-biologic DMARD use; LS Mean Treatment Difference = -0.40, 95% CI 2-sided [-0.62 to -0.17], Standard Error of Mean 0.12 — Methotrexate Monotherapy is the reference

18. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire- Disability Index (HAQ-DI) at Week 24
Description: The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire consisting of 20 questions referring in 8 functional areas: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and usual activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task are summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. Negative mean changes from Baseline in the overall score indicate improvement in functional ability.
Time Frame: Baseline and week 24
Population: All randomized participants with available data
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 252 | 258 | 257
units on a scale | -0.412 (0.036) | -0.444 (0.035) | -0.468 (0.038)
Statistical Analysis 1: Comparison: Methotrexate Monotherapy vs Etanercept + Methotrexate; Test type: Superiority; p = 0.34, ANCOVA — P-value is unadjusted and considered descriptive; ANCOVA model adjusted for baseline BMI status (≤ 30 kg/m² or >30 kg/m²) and prior non-biologic DMARD use; LS Mean Treatment Difference = -0.05, 95% CI 2-sided [-0.15 to 0.05], Standard Error of Mean 0.05 — Methotrexate Monotherapy is the reference
Statistical Analysis 2: Comparison: Methotrexate Monotherapy vs Etanercept Monotherapy; Test type: Superiority; p = 0.67, ANCOVA — P-value is unadjusted and considered descriptive; ANCOVA model adjusted for baseline BMI status (≤ 30 kg/m² or > 30 kg/m²) and prior non-biologic DMARD use; LS Mean Treatment Difference = -0.02, 95% CI 2-sided [-0.12 to 0.08], Standard Error of Mean 0.05 — Methotrexate Monotherapy is the reference

19. Secondary Outcome: Change From Baseline in Medical Outcomes Health Survey Short Form 36 Items Version 2 (SF-36 v2) at Week 24
Description: The SF-36 is a health-related survey that assesses participant's quality of life and consists of 36 questions covering 8 health domains. Two summary component scores are calculated: mental component summary score (MCS) and physical component summary score (PCS). The MCS consists of social functioning, vitality, mental health, and role-emotional scales and the PCS consists of physical functioning, bodily pain, role-physical, and general health scales. Each domain is scored by summing the individual items and transforming the scores into a 0 to 100 scale with higher scores indicating better health status or functioning.
Time Frame: Baseline and week 24
Population: All randomized participants with available data
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 253 | 256 | 257
units on a scale
  Physical Component Summary | 5.952 (0.550) | 7.808 (0.546) | 8.011 (0.598)
  Mental Component Summary | 3.259 (0.589) | 2.835 (0.624) | 3.321 (0.572)
Statistical Analysis 1: Comparison: Methotrexate Monotherapy vs Etanercept + Methotrexate; Analysis of change from baseline in Physical Component Summary at week 24; Test type: Superiority; p = 0.015, ANCOVA — P-value is unadjusted and considered descriptive; ANCOVA model adjusted for baseline BMI status (≤ 30 kg/m² or >30 kg/m²) and prior non-biologic DMARD use; LS Mean Treatment Difference = 1.94, 95% CI 2-sided [0.37 to 3.51], Standard Error of Mean 0.80 — Methotrexate Monotherapy is the reference
Statistical Analysis 2: Comparison: Methotrexate Monotherapy vs Etanercept Monotherapy; Analysis of change from baseline in Physical Component Summary at week 24; Test type: Superiority; p = 0.033, ANCOVA — P-value is unadjusted and considered descriptive; ANCOVA model adjusted for baseline BMI status (≤ 30 kg/m² or > 30 kg/m²) and prior non-biologic DMARD use; LS Mean Treatment Difference = 1.71, 95% CI 2-sided [0.13 to 3.28], Standard Error of Mean 0.80 — Methotrexate Monotherapy is the reference
Statistical Analysis 3: Comparison: Methotrexate Monotherapy vs Etanercept + Methotrexate; Analysis of change from baseline in Mental Component Summary at week 24; Test type: Superiority; p = 0.97, ANCOVA — P-value is unadjusted and considered descriptive; ANCOVA model adjusted for baseline BMI status (≤ 30 kg/m² or > 30 kg/m²) and prior non-biologic DMARD use; LS Mean Treatment Difference = -0.03, 95% CI 2-sided [-1.69 to 1.63], Standard Error of Mean 0.84 — Methotrexate Monotherapy is the reference
Statistical Analysis 4: Comparison: Methotrexate Monotherapy vs Etanercept Monotherapy; Analysis of change from baseline in Mental Component Summary at week 24; Test type: Superiority; p = 0.56, ANCOVA — P-value is unadjusted and considered descriptive; ANCOVA model adjusted for baseline BMI status (≤ 30 kg/m² or > 30 kg/m²) and prior non-biologic DMARD use; LS Mean Treatment Difference = -0.50, 95% CI 2-sided [-2.16 to 1.16], Standard Error of Mean 0.85 — Methotrexate Monotherapy is the reference

20. Secondary Outcome: Change From Baseline in Modified Nail Psoriasis Severity Index (mNAPSI) at Week 24
Description: The modified NAPSI scale is a grading system for nail psoriasis that incorporates the following 7 clinical features:
  * pitting (scores 0-3, depending on the number of pits)
  * nail plate crumbling (scores 0-3, depending on the % of nail involvement)
  * onycholysis and oil drop dyschromia (scores 0-3, depending on the % of nail involvement)
  * leukonychia (0 = absent, 1 = present)
  * red spots in lunula (0 = absent, 1 = present)
  * nail bed hyperkeratosis (0 = absent, 1 = present)
  * splinter hemorrhages (0 = absent, 1 = present)
  In participants with fingernails involved with psoriasis, each fingernail was scored at baseline to determine the worst fingernail (ie, the fingernail with the highest mNAPSI score). This fingernail was followed for the remainder of the study.
  mNAPSI scores range from 0-13 where higher scores represent worse nail disease.
Time Frame: Baseline and week 24
Population: Randomized participants with non-zero mNAPSI score at baseline and available data at week 24
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 121 | 115 | 123
units on a scale | -1.1 (0.2) | -1.5 (0.2) | -1.7 (0.2)
Statistical Analysis 1: Comparison: Methotrexate Monotherapy vs Etanercept + Methotrexate; Test type: Superiority; p = 0.020, ANCOVA — P-value is unadjusted and considered descriptive; ANCOVA model adjusted for baseline BMI status (≤ 30 kg/m² or >30 kg/m²) and prior non-biologic DMARD use; LS Mean Treatment Difference = -0.56, 95% CI 2-sided [-1.03 to -0.09], Standard Error of Mean 0.24 — Methotrexate Monotherapy is the reference
Statistical Analysis 2: Comparison: Methotrexate Monotherapy vs Etanercept Monotherapy; Test type: Superiority; p = 0.10, ANCOVA — P-value is unadjusted and considered descriptive; ANCOVA model adjusted for baseline BMI status (≤ 30 kg/m² or > 30 kg/m²) and prior non-biologic DMARD use; LS Mean Treatment Difference = -0.40, 95% CI 2-sided [-0.88 to 0.08], Standard Error of Mean 0.24 — Methotrexate Monotherapy is the reference

21. Secondary Outcome: Percentage of Participants With Clear mNAPSI at Week 24
Description: The modified NAPSI scale is a grading system for nail psoriasis that incorporates the following 7 clinical features:
  * pitting (scores 0-3, depending on the number of pits)
  * nail plate crumbling (scores 0-3, depending on the % of nail involvement)
  * onycholysis and oil drop dyschromia (scores 0-3, depending on the % of nail involvement)
  * leukonychia (0 = absent, 1 = present)
  * red spots in lunula (0 = absent, 1 = present)
  * nail bed hyperkeratosis (0 = absent, 1 = present)
  * splinter hemorrhages (0 = absent, 1 = present)
  In participants with fingernails involved with psoriasis, each fingernail was scored at baseline to determine the worst fingernail (ie, the fingernail with the highest mNAPSI score). This fingernail was followed for the remainder of the study.
  mNAPSI scores range from 0-13 where higher scores represent worse nail disease. Clear mNAPSI is defined as a score = 0.
Time Frame: Baseline and week 24
Population: Randomized participants with non-zero mNAPSI score at baseline and available data at week 24
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 121 | 115 | 123
percentage of participants | 0.0 | 0.0 | 0.0

22. Secondary Outcome: Change From Baseline in Leeds Dactylitis Index (LDI) at Week 24
Description: The Leeds dactylitis index quantitatively measures dactylitis using the circumference of involved digits and control digits and tenderness of involved digits. Digits affected by dactylitis are defined as those with a 10% difference in the ratio of circumference of the affected digit to the contralateral digit. The control digit is either the contralateral digit (digit on opposite hand or foot), or if the contralateral digit is also affected, values from a standard reference table. Tenderness of affected digits is assessed on a scale from 0 [none] to 3 [worst]. The ratio of circumference between an affected digit and the control digit is multiplied by the tenderness score for the affected digit. The results from each involved digit are summed to provide the final LDI. A higher LDI indicates worse dactylitis.
Time Frame: Baseline and week 24
Population: Randomized participants with non-zero LDI score at baseline and available data at week 24
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 89 | 89 | 87
units on a scale | -128.80 (26.76) | -119.09 (20.66) | -110.15 (22.70)
Statistical Analysis 1: Comparison: Methotrexate Monotherapy vs Etanercept + Methotrexate; Test type: Superiority; p = 0.68, ANCOVA — P-value is unadjusted and considered descriptive; ANCOVA model adjusted for baseline BMI status (≤ 30 kg/m² or >30 kg/m²) and prior non-biologic DMARD use; LS Mean Treatment Difference = 13.92, 95% CI 2-sided [-51.52 to 79.36], Standard Error of Mean 33.23 — Methotrexate Monotherapy is the reference
Statistical Analysis 2: Comparison: Methotrexate Monotherapy vs Etanercept Monotherapy; Test type: Superiority; p = 0.85, ANCOVA — P-value is unadjusted and considered descriptive; ANCOVA model adjusted for baseline BMI status (≤ 30 kg/m² or > 30 kg/m²) and prior non-biologic DMARD use; LS Mean Treatment Difference = 6.34, 95% CI 2-sided [-58.75 to 71.42], Standard Error of Mean 33.05 — Methotrexate Monotherapy is the reference

23. Secondary Outcome: Percentage of Participants With Clear LDI at Week 24
Description: The Leeds dactylitis index quantitatively measures dactylitis using the circumference of involved digits and control digits and tenderness of involved digits. Digits affected by dactylitis are defined as those with a 10% difference in the ratio of circumference of the affected digit to the contralateral digit. The control digit is either the contralateral digit (digit on opposite hand or foot), or if the contralateral digit is also affected, values from a standard reference table. Tenderness of affected digits is assessed on a scale from 0 [none] to 3 [worst]. The ratio of circumference between an affected digit and the control digit is multiplied by the tenderness score for the affected digit. The results from each involved digit are summed to provide the final LDI. A higher LDI indicates worse dactylitis.
  Clear LDI is defined as a score = 0.
Time Frame: Baseline and week 24
Population: Randomized participants with non-zero LDI score at baseline and available data at week 24
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 89 | 89 | 87
percentage of participants | 65.2 | 76.4 | 79.3
Statistical Analysis 1: Comparison: Methotrexate Monotherapy vs Etanercept + Methotrexate; Test type: Superiority; p = 0.057, Cochran-Mantel-Haenszel — P-value is unadjusted and considered descriptive; [statistical method as in outcome 1, analysis 1]; Treatment Difference = 12.9, 95% CI 2-sided [-0.4 to 26.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Methotrexate Monotherapy vs Etanercept Monotherapy; Test type: Superiority; p = 0.12, Cochran-Mantel-Haenszel — P-value is unadjusted and considered descriptive; [statistical method as in outcome 1, analysis 1]; Treatment Difference = 10.9, 95% CI 2-sided [-2.5 to 24.4] — [estimate comment as in outcome 1, analysis 1]

24. Secondary Outcome: Change From Baseline in Spondyloarthritis Research Consortium of Canada (SPARCC) Enthesitis Index at Week 24
Description: The SPARCC enthesitis index assesses enthesitis at 18 sites for palpitation with a resultant total score of 0 to 16 (for scoring purposes, the inferior patella and tibial tuberosity are considered 1 site because of their anatomical proximity). Tenderness at each site is quantified on a dichotomous basis (0 = non-tender, 1 = tender). Entheses assessed are medial epicondyle (left and right), lateral epicondyle (left and right), supraspinatus insertion into greater tuberosity of humerus (left and right), greater trochanter (left and right), quadriceps insertion into superior border of patella (left and right), patellar ligament insertion into inferior pole of patella or tibial tubercle (left and right), Achilles tendon insertion into calcaneum (left and right), plantar fascia insertion into calcaneum (left and right). A higher count represents greater enthesitis burden.
Time Frame: Baseline and week 24
Population: Randomized participants with non-zero SPARCC enthesitis index score at baseline and available data at week 24
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 167 | 173 | 179
units on a scale | -3.1 (0.3) | -3.0 (0.3) | -2.9 (0.3)
Statistical Analysis 1: Comparison: Methotrexate Monotherapy vs Etanercept + Methotrexate; Test type: Superiority; p = 0.70, ANCOVA — P-value is unadjusted and considered descriptive; ANCOVA model adjusted for baseline BMI status (≤ 30 kg/m² or >30 kg/m²) and prior non-biologic DMARD use; LS Mean Treatment Difference = 0.16, 95% CI 2-sided [-0.66 to 0.98], Standard Error of Mean 0.42 — Methotrexate Monotherapy is the reference
Statistical Analysis 2: Comparison: Methotrexate Monotherapy vs Etanercept Monotherapy; Test type: Superiority; p = 0.93, ANCOVA — P-value is unadjusted and considered descriptive; ANCOVA model adjusted for baseline BMI status (≤ 30 kg/m² or > 30 kg/m²) and prior non-biologic DMARD use; LS Mean Treatment Difference = 0.04, 95% CI 2-sided [-0.79 to 0.86], Standard Error of Mean 0.42 — Methotrexate Monotherapy is the reference

25. Secondary Outcome: Percentage of Participants With Clear SPARCC Enthesitis Index Score at Week 24
Description: The SPARCC enthesitis index assesses enthesitis at 18 sites for palpitation with a resultant total score of 0 to 16 (for scoring purposes, the inferior patella and tibial tuberosity are considered 1 site because of their anatomical proximity). Tenderness at each site is quantified on a dichotomous basis (0 = non-tender, 1 = tender). Entheses assessed are medial epicondyle (left and right), lateral epicondyle (left and right), supraspinatus insertion into greater tuberosity of humerus (left and right), greater trochanter (left and right), quadriceps insertion into superior border of patella (left and right), patellar ligament insertion into inferior pole of patella or tibial tubercle (left and right), Achilles tendon insertion into calcaneum (left and right), plantar fascia insertion into calcaneum (left and right). A higher count represents greater enthesitis burden.
  Clear SPARCC enthesitis is defined as a score = 0.
Time Frame: Baseline and week 24
Population: Randomized participants with non-zero SPARCC enthesitis index score at baseline and available data at week 24
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 167 | 173 | 179
percentage of participants | 43.1 | 52.6 | 47.8
Statistical Analysis 1: Comparison: Methotrexate Monotherapy vs Etanercept + Methotrexate; Test type: Superiority; p = 0.55, Cochran-Mantel-Haenszel — P-value is unadjusted and considered descriptive; [statistical method as in outcome 1, analysis 1]; Treatment Difference = 3.2, 95% CI 2-sided [-7.3 to 13.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Methotrexate Monotherapy vs Etanercept Monotherapy; Test type: Superiority; p = 0.11, Cochran-Mantel-Haenszel — P-value is unadjusted and considered descriptive; [statistical method as in outcome 1, analysis 1]; Treatment Difference = 8.8, 95% CI 2-sided [-1.9 to 19.4] — [estimate comment as in outcome 1, analysis 1]

26. Secondary Outcome: Percent Improvement From Baseline in the Percentage of Body Surface Area (BSA) Involved in Psoriasis at Week 24
Description: The physician's assessment of the percentage of the participant's total body surface area involved with psoriasis.
  Percent improvement from baseline = (Baseline Value - Post-baseline Value) / Baseline * 100
Time Frame: Baseline and week 24
Population: Randomized participants with ≥ 3% body surface area (BSA) psoriasis involvement at baseline and available data.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 179 | 166 | 163
percent change | 66.12 (2.76) | 69.80 (2.73) | 75.53 (3.71)
Statistical Analysis 1: Comparison: Methotrexate Monotherapy vs Etanercept + Methotrexate; Test type: Superiority; p = 0.031, ANCOVA — P-value is unadjusted and considered descriptive; ANCOVA model adjusted for baseline BMI status (≤ 30 kg/m² or >30 kg/m²) and prior non-biologic DMARD use; LS Mean Treatment Difference = 9.36, 95% CI 2-sided [0.85 to 17.87], Standard Error of Mean 4.33 — Methotrexate Monotherapy is the reference
Statistical Analysis 2: Comparison: Methotrexate Monotherapy vs Etanercept Monotherapy; Test type: Superiority; p = 0.49, ANCOVA — P-value is unadjusted and considered descriptive; ANCOVA model adjusted for baseline BMI status (≤ 30 kg/m² or > 30 kg/m²) and prior non-biologic DMARD use; LS Mean Treatment Difference = 3.02, 95% CI 2-sided [-5.49 to 11.54], Standard Error of Mean 4.33 — Methotrexate Monotherapy is the reference

27. Secondary Outcome: Percent Improvement From Baseline in the Percentage of Body Surface Area (BSA) Involved in Psoriasis by Baseline BSA Involvement Subgroups
Description: as for outcome 26
Time Frame: Baseline and week 24
Population: Randomized participants with available BSA data
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 254 | 259 | 259
percent change
  < 3% BSA involvement at baseline: number analyzed (Participants) | 75 | 93 | 96
  < 3% BSA involvement at baseline | -24.49 (46.71) | -92.18 (108.54) | 17.66 (51.97)
  ≥ 3% to < 10% BSA involvement at baseline: number analyzed (Participants) | 87 | 75 | 77
  ≥ 3% to < 10% BSA involvement at baseline | 66.61 (4.18) | 64.42 (4.43) | 68.76 (7.26)
  ≥ 10% BSA involvement at baseline: number analyzed (Participants) | 92 | 91 | 86
  ≥ 10% BSA involvement at baseline | 65.66 (3.66) | 74.23 (3.32) | 81.61 (2.55)
Statistical Analysis 1: Comparison: Methotrexate Monotherapy vs Etanercept + Methotrexate; Analysis of percent improvement from baseline in the percentage of BSA involved in psoriasis in the subgroup of participants with ≥ 10% BSA involvement at baseline; Test type: Superiority; p < 0.001, ANCOVA — P-value is unadjusted and considered descriptive; ANCOVA model adjusted for baseline BMI status (≤ 30 kg/m² or > 30 kg/m²) and prior non-biologic DMARD use; LS Mean Treatment Difference = 15.95, 95% CI 2-sided [6.99 to 24.90], Standard Error of Mean 4.55 — Methotrexate Monotherapy is the reference
Statistical Analysis 2: Comparison: Methotrexate Monotherapy vs Etanercept Monotherapy; [analysis description as in outcome 27, analysis 1]; Test type: Superiority; p = 0.12, ANCOVA — P-value is unadjusted and considered descriptive; ANCOVA model adjusted for baseline BMI status (≤ 30 kg/m² or > 30 kg/m²) and prior non-biologic DMARD use; LS Mean Treatment Difference = 6.97, 95% CI 2-sided [-1.89 to 15.83], Standard Error of Mean 4.50 — Methotrexate Monotherapy is the reference

28. Secondary Outcome: Static Physician Global Assessment (sPGA) at Week 24
Description: The static Physician Global Assessment of psoriasis (sPGA) evaluates the physician's global assessment of the participant's psoriasis based on severity of induration, scaling, and erythema. The sPGA is assessed on a scale from 0 to 5:
  0 = clear (no evidence of plaque elevation, erythema or scaling)
  1. = almost clear (minimal plaque elevation, erythema or scaling)
  2. = mild (mild plaque elevation or scaling, light red coloration)
  3. = moderate (moderate plaque elevation, scaling, light red coloration)
  4. = marked (marked plaque elevation, thick, non-tenacious scale predominates, bright red coloration)
  5. = severe (severe plaque elevation, very thick tenacious scaling, dusky to deep red coloration).
Time Frame: Week 24
Population: Randomized participants with ≥ 3% body surface area (BSA) psoriasis involvement at baseline and available sPGA data.
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 178 | 166 | 161
Participants
  0 (clear) | 38 | 36 | 63
  1 (almost clear) | 80 | 84 | 62
  2 (mild) | 34 | 28 | 25
  3 (moderate) | 22 | 12 | 10
  4 (marked) | 3 | 6 | 1
  5 (severe) | 1 | 0 | 0

29. Secondary Outcome: Static Physician Global Assessment (sPGA) at Week 24 by Baseline BSA Involvement Subgroups
Description: as for outcome 28
Time Frame: Week 24
Population: Randomized participants with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 253 | 258 | 257
Participants
  < 3% BSA involvement at baseline: number analyzed (Participants) | 75 | 92 | 96
  < 3% BSA involvement at baseline: 0 (clear) | 26 | 29 | 52
  < 3% BSA involvement at baseline: 1 (almost clear) | 28 | 37 | 32
  < 3% BSA involvement at baseline: 2 (mild) | 15 | 19 | 9
  < 3% BSA involvement at baseline: 3 (moderate) | 4 | 6 | 3
  < 3% BSA involvement at baseline: 4 (marked) | 2 | 1 | 0
  < 3% BSA involvement at baseline: 5 (severe) | 0 | 0 | 0
  ≥ 3% to < 10% BSA involvement at baseline: number analyzed (Participants) | 87 | 75 | 76
  ≥ 3% to < 10% BSA involvement at baseline: 0 (clear) | 23 | 16 | 35
  ≥ 3% to < 10% BSA involvement at baseline: 1 (almost clear) | 41 | 32 | 23
  ≥ 3% to < 10% BSA involvement at baseline: 2 (mild) | 13 | 18 | 12
  ≥ 3% to < 10% BSA involvement at baseline: 3 (moderate) | 10 | 7 | 5
  ≥ 3% to < 10% BSA involvement at baseline: 4 (marked) | 0 | 2 | 1
  ≥ 3% to < 10% BSA involvement at baseline: 5 (severe) | 0 | 0 | 0
  ≥ 10% BSA involvement at baseline: number analyzed (Participants) | 91 | 91 | 85
  ≥ 10% BSA involvement at baseline: 0 (clear) | 15 | 20 | 28
  ≥ 10% BSA involvement at baseline: 1 (almost clear) | 39 | 52 | 39
  ≥ 10% BSA involvement at baseline: 2 (mild) | 21 | 10 | 13
  ≥ 10% BSA involvement at baseline: 3 (moderate) | 12 | 5 | 5
  ≥ 10% BSA involvement at baseline: 4 (marked) | 3 | 4 | 0
  ≥ 10% BSA involvement at baseline: 5 (severe) | 1 | 0 | 0

30. Secondary Outcome: Mean Static Physician Global Assessment (sPGA) Score at Week 24
Description: as for outcome 28
Time Frame: Week 24
Population: Randomized participants with ≥ 3% body surface area (BSA) psoriasis involvement at baseline and available sPGA data.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 178 | 166 | 161
units on a scale | 1.3 (0.1) | 1.2 (0.1) | 0.9 (0.1)

31. Secondary Outcome: Mean Static Physician Global Assessment (sPGA) Score at Week 24 by Baseline BSA Involvement Subgroups
Description: as for outcome 28
Time Frame: Week 24
Population: Randomized participants with available data
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 253 | 258 | 257
units on a scale
  < 3% BSA involvement at baseline: number analyzed (Participants) | 75 | 92 | 96
  < 3% BSA involvement at baseline | 1.0 (0.1) | 1.1 (0.1) | 0.6 (0.1)
  ≥ 3% to < 10% BSA involvement at baseline: number analyzed (Participants) | 87 | 75 | 76
  ≥ 3% to < 10% BSA involvement at baseline | 1.1 (0.1) | 1.3 (0.1) | 0.9 (0.1)
  ≥ 10% BSA involvement at baseline: number analyzed (Participants) | 91 | 91 | 85
  ≥ 10% BSA involvement at baseline | 1.5 (0.1) | 1.1 (0.1) | 0.9 (0.1)

32. Secondary Outcome: Percentage of Participants With an sPGA Score of 0 (Clear) or 1 (Almost Clear) at Week 24
Description: as for outcome 28
Time Frame: Week 24
Population: Randomized participants with ≥ 3% body surface area (BSA) psoriasis involvement at baseline and available sPGA data.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 178 | 166 | 161
percentage of participants | 66.3 | 72.3 | 77.6
Statistical Analysis 1: Comparison: Methotrexate Monotherapy vs Etanercept + Methotrexate; Test type: Superiority; p = 0.019, Cochran-Mantel-Haenszel — P-value is unadjusted and considered descriptive; [statistical method as in outcome 1, analysis 1]; Treatment Difference = 11.4, 95% CI 2-sided [2.0 to 20.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Methotrexate Monotherapy vs Etanercept Monotherapy; Test type: Superiority; p = 0.40, Cochran-Mantel-Haenszel — P-value is unadjusted and considered descriptive; [statistical method as in outcome 1, analysis 1]; Treatment Difference = 4.2, 95% CI 2-sided [-5.6 to 14.0] — [estimate comment as in outcome 1, analysis 1]

33. Secondary Outcome: Percentage of Participants With an sPGA Score of 0 (Clear) or 1 (Almost Clear) at Week 24 by Baseline BSA Involvement Subgroups
Description: as for outcome 28
Time Frame: Week 24
Population: Randomized participants with available data
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 253 | 258 | 257
percentage of participants
  < 3% BSA involvement at baseline: number analyzed (Participants) | 75 | 92 | 96
  < 3% BSA involvement at baseline | 72.0 | 71.7 | 87.5
  ≥ 3% to < 10% BSA involvement at baseline: number analyzed (Participants) | 87 | 75 | 76
  ≥ 3% to < 10% BSA involvement at baseline | 73.6 | 64.0 | 76.3
  ≥ 10% BSA involvement at baseline: number analyzed (Participants) | 91 | 91 | 85
  ≥ 10% BSA involvement at baseline | 59.3 | 79.1 | 78.8
Statistical Analysis 1: Comparison: Methotrexate Monotherapy vs Etanercept + Methotrexate; Analysis of percentage of participants with an sPGA of 0 or 1 at Week 24 in participants with baseline BSA involvement with psoriasis ≥ 10%; Test type: Superiority; p = 0.004, Cochran-Mantel-Haenszel — P-value is unadjusted and considered descriptive; [statistical method as in outcome 1, analysis 1]; Treatment Difference = 20.1, 95% CI 2-sided [6.8 to 33.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Methotrexate Monotherapy vs Etanercept Monotherapy; [analysis description as in outcome 33, analysis 1]; Test type: Superiority; p = 0.012, Cochran-Mantel-Haenszel — P-value is unadjusted and considered descriptive; [statistical method as in outcome 1, analysis 1]; Treatment Difference = 17.1, 95% CI 2-sided [4.0 to 30.2] — [estimate comment as in outcome 1, analysis 1]

34. Secondary Outcome: Percentage of Participants With at Least a 1 Grade Improvement in sPGA From Baseline at Week 24
Description: as for outcome 28
Time Frame: Baseline and week 24
Population: Randomized participants with ≥ 3% body surface area (BSA) psoriasis involvement at baseline and available sPGA data.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 177 | 166 | 161
percentage of participants | 29.9 | 28.9 | 18.0

35. Secondary Outcome: Percentage of Participants With at Least a 1 Grade Improvement in sPGA From Baseline at Week 24 by Baseline BSA Involvement Subgroups
Description: as for outcome 28
Time Frame: Baseline and week 24
Population: Randomized participants with available data
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 250 | 258 | 257
percentage of participants
  < 3% BSA involvement at baseline: number analyzed (Participants) | 73 | 92 | 96
  < 3% BSA involvement at baseline | 37.0 | 44.6 | 43.8
  ≥ 3% to < 10% BSA involvement at baseline: number analyzed (Participants) | 86 | 75 | 76
  ≥ 3% to < 10% BSA involvement at baseline | 27.9 | 38.7 | 21.1
  ≥ 10% BSA involvement at baseline: number analyzed (Participants) | 91 | 91 | 85
  ≥ 10% BSA involvement at baseline | 31.9 | 20.9 | 15.3

36. Secondary Outcome: Percentage of Participants With at Least a 2 Grade Improvement in sPGA From Baseline at Week 24
Description: as for outcome 28
Time Frame: Baseline and week 24
Population: Randomized participants with ≥ 3% body surface area (BSA) psoriasis involvement at baseline and available sPGA data.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 177 | 166 | 161
percentage of participants | 30.5 | 28.9 | 35.4

37. Secondary Outcome: Percentage of Participants With at Least a 2 Grade Improvement in sPGA From Baseline at Week 24 by Baseline BSA Involvement Subgroups
Description: as for outcome 28
Time Frame: Baseline and week 24
Population: Randomized participants with available data
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
Number analyzed (Participants) | 250 | 258 | 257
percentage of participants
  < 3% BSA involvement at baseline: number analyzed (Participants) | 73 | 92 | 96
  < 3% BSA involvement at baseline | 15.1 | 20.7 | 30.2
  ≥ 3% to < 10% BSA involvement at baseline: number analyzed (Participants) | 86 | 75 | 76
  ≥ 3% to < 10% BSA involvement at baseline | 34.9 | 25.3 | 32.9
  ≥ 10% BSA involvement at baseline: number analyzed (Participants) | 91 | 91 | 85
  ≥ 10% BSA involvement at baseline | 26.4 | 31.9 | 37.6

ADVERSE EVENTS:
Time Frame: 48-week treatment period plus 30-day safety follow-up
Description: Two participants randomized to the Etanercept Monotherapy arm also received methotrexate in error, so are counted in the Etanercept + Methotrexate group for safety.
  Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Methotrexate Monotherapy | Etanercept Monotherapy | Etanercept + Methotrexate
All-Cause Mortality (participants affected / at risk) | 0/282 | 0/282 | 0/284
Serious Adverse Events (participants affected / at risk) | 16/282 | 19/282 | 17/284
Other Adverse Events (participants affected / at risk) | 210/282 | 185/282 | 214/284
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methotrexate Monotherapy (N=282) | Etanercept Monotherapy (N=282) | Etanercept + Methotrexate (N=284)
Acute myocardial infarction (Cardiac disorders) | 2 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0
Supraventricular tachyarrhythmia (Cardiac disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 2
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0 | 0
Acute pulmonary histoplasmosis (Infections and infestations) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 2
Bronchitis (Infections and infestations) | 0 | 2 | 1
Cellulitis (Infections and infestations) | 0 | 2 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Necrotising fasciitis streptococcal (Infections and infestations) | 0 | 1 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1
Pneumonia necrotising (Infections and infestations) | 0 | 0 | 1
Post procedural sepsis (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 1
Foreign body (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Migraine (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0
Radiculopathy (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 2 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Spinal fusion surgery (Surgical and medical procedures) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methotrexate Monotherapy (N=282) | Etanercept Monotherapy (N=282) | Etanercept + Methotrexate (N=284)
Anaemia (Blood and lymphatic system disorders) | 4 | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 1 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Cor pulmonale (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0
Extrasystoles (Cardiac disorders) | 1 | 0 | 0
Left ventricular hypertrophy (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 2
Pericarditis (Cardiac disorders) | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 1
Kidney malformation (Congenital, familial and genetic disorders) | 0 | 0 | 1
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 2 | 1 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 5
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 1 | 2
Thyroid mass (Endocrine disorders) | 0 | 0 | 1
Abnormal sensation in eye (Eye disorders) | 0 | 1 | 0
Blepharitis (Eye disorders) | 1 | 0 | 0
Blindness unilateral (Eye disorders) | 1 | 0 | 0
Diabetic retinopathy (Eye disorders) | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 2
Eye irritation (Eye disorders) | 0 | 1 | 1
Iridocyclitis (Eye disorders) | 0 | 0 | 1
Myopia (Eye disorders) | 0 | 1 | 1
Pterygium (Eye disorders) | 0 | 1 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1
Vitreous detachment (Eye disorders) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 2 | 5
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 3 | 5
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 7 | 7 | 6
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 2 | 2 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 1 | 3
Dental caries (Gastrointestinal disorders) | 1 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 17 | 13 | 14
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 5 | 2 | 3
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Gastric disorder (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 4 | 3 | 2
Gastritis erosive (Gastrointestinal disorders) | 0 | 1 | 0
Gastroduodenitis (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 2 | 4
Glossodynia (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 2 | 1 | 2
Mucous stools (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 37 | 18 | 41
Odynophagia (Gastrointestinal disorders) | 1 | 2 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatic disorder (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 0 | 1
Toothache (Gastrointestinal disorders) | 5 | 0 | 4
Vomiting (Gastrointestinal disorders) | 15 | 7 | 10
Administration site rash (General disorders) | 0 | 0 | 1
Adverse drug reaction (General disorders) | 0 | 0 | 1
Application site bruise (General disorders) | 0 | 1 | 0
Asthenia (General disorders) | 2 | 1 | 3
Chest discomfort (General disorders) | 0 | 0 | 1
Chest pain (General disorders) | 2 | 0 | 2
Chills (General disorders) | 0 | 0 | 2
Cyst (General disorders) | 0 | 1 | 0
Drug intolerance (General disorders) | 1 | 0 | 1
Early satiety (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 8 | 5 | 10
General physical health deterioration (General disorders) | 0 | 1 | 0
Influenza like illness (General disorders) | 7 | 2 | 3
Injection site bruising (General disorders) | 2 | 1 | 2
Injection site erythema (General disorders) | 1 | 5 | 5
Injection site extravasation (General disorders) | 0 | 2 | 0
Injection site haematoma (General disorders) | 0 | 1 | 0
Injection site inflammation (General disorders) | 0 | 1 | 0
Injection site irritation (General disorders) | 0 | 1 | 0
Injection site oedema (General disorders) | 0 | 1 | 0
Injection site pain (General disorders) | 0 | 2 | 3
Injection site pruritus (General disorders) | 1 | 0 | 1
Injection site rash (General disorders) | 1 | 4 | 4
Injection site reaction (General disorders) | 1 | 5 | 8
Malaise (General disorders) | 1 | 2 | 2
Nodule (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 3 | 2 | 2
Oedema peripheral (General disorders) | 1 | 5 | 0
Pain (General disorders) | 1 | 3 | 1
Peripheral swelling (General disorders) | 2 | 1 | 0
Puncture site erythema (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 5 | 3 | 6
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 2
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 0
Gallbladder disorder (Hepatobiliary disorders) | 0 | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 2 | 3 | 1
Hepatobiliary disease (Hepatobiliary disorders) | 1 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 1 | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0 | 0
Allergy to arthropod sting (Immune system disorders) | 0 | 1 | 1
Allergy to plants (Immune system disorders) | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 2 | 2
Abscess limb (Infections and infestations) | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 1 | 3 | 0
Adenoviral upper respiratory infection (Infections and infestations) | 1 | 0 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1
Body tinea (Infections and infestations) | 0 | 2 | 0
Bronchitis (Infections and infestations) | 9 | 12 | 18
Bronchitis viral (Infections and infestations) | 0 | 1 | 0
Candida infection (Infections and infestations) | 1 | 0 | 0
Carbuncle (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 5
Chorioretinitis (Infections and infestations) | 0 | 1 | 0
Chronic sinusitis (Infections and infestations) | 1 | 1 | 0
Chronic tonsillitis (Infections and infestations) | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 2 | 0 | 1
Cystitis (Infections and infestations) | 0 | 1 | 2
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Ear infection (Infections and infestations) | 3 | 1 | 2
Folliculitis (Infections and infestations) | 2 | 0 | 2
Fungal infection (Infections and infestations) | 0 | 2 | 0
Furuncle (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 3 | 4 | 8
Gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 1 | 3
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0
Gingivitis (Infections and infestations) | 2 | 0 | 0
Helicobacter infection (Infections and infestations) | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0 | 0
Herpes virus infection (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 2 | 2 | 1
Impetigo (Infections and infestations) | 0 | 1 | 0
Infected bite (Infections and infestations) | 0 | 1 | 1
Infected cyst (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 9 | 7 | 8
Laryngitis (Infections and infestations) | 3 | 0 | 1
Laryngitis viral (Infections and infestations) | 0 | 0 | 1
Localised infection (Infections and infestations) | 1 | 1 | 2
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Lymph node abscess (Infections and infestations) | 0 | 0 | 1
Nail bed infection (Infections and infestations) | 2 | 0 | 0
Nasal herpes (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 22 | 21 | 27
Onychomycosis (Infections and infestations) | 1 | 0 | 0
Ophthalmic herpes simplex (Infections and infestations) | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0
Oral herpes (Infections and infestations) | 4 | 1 | 3
Oral infection (Infections and infestations) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 1
Otitis media (Infections and infestations) | 1 | 1 | 0
Paronychia (Infections and infestations) | 1 | 0 | 1
Periodontitis (Infections and infestations) | 0 | 2 | 0
Pertussis (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 2 | 1 | 5
Pharyngitis bacterial (Infections and infestations) | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 2 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1
Post procedural pneumonia (Infections and infestations) | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
Pulpitis dental (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 3 | 3 | 5
Respiratory tract infection viral (Infections and infestations) | 3 | 5 | 1
Rhinitis (Infections and infestations) | 4 | 4 | 2
Rhinovirus infection (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 8 | 11 | 8
Sinusitis bacterial (Infections and infestations) | 1 | 0 | 0
Skin candida (Infections and infestations) | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 1
Tinea versicolour (Infections and infestations) | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 2 | 1 | 3
Tooth abscess (Infections and infestations) | 2 | 3 | 3
Tooth infection (Infections and infestations) | 2 | 3 | 2
Tracheitis (Infections and infestations) | 0 | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 21 | 18 | 23
Urinary tract infection (Infections and infestations) | 4 | 4 | 1
Vaginal infection (Infections and infestations) | 0 | 0 | 2
Viral infection (Infections and infestations) | 3 | 4 | 3
Viral pharyngitis (Infections and infestations) | 1 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 2 | 1
Wound infection (Infections and infestations) | 0 | 1 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 0 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 3 | 1 | 3
Dental restoration failure (Injury, poisoning and procedural complications) | 0 | 0 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 3 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 2 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Foreign body in eye (Injury, poisoning and procedural complications) | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 2 | 3
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 3 | 4
Limb injury (Injury, poisoning and procedural complications) | 1 | 1 | 1
Lip injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 3 | 2 | 2
Nail avulsion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tooth avulsion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1 | 2
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 1 | 0
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 2 | 1
Alanine aminotransferase increased (Investigations) | 9 | 4 | 13
Aspartate aminotransferase increased (Investigations) | 7 | 3 | 6
Blood bilirubin abnormal (Investigations) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Blood cholesterol increased (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0
Blood glucose abnormal (Investigations) | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1
Blood triglycerides abnormal (Investigations) | 0 | 0 | 1
Blood urea increased (Investigations) | 1 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 1
Body temperature increased (Investigations) | 1 | 0 | 1
Borrelia test positive (Investigations) | 1 | 0 | 0
Endoscopy gastrointestinal (Investigations) | 0 | 1 | 0
Hepatic enzyme abnormal (Investigations) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 6 | 2 | 2
Liver function test abnormal (Investigations) | 2 | 0 | 2
Liver function test increased (Investigations) | 1 | 0 | 0
Low density lipoprotein increased (Investigations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0
Precancerous cells present (Investigations) | 0 | 0 | 1
Prostatic specific antigen abnormal (Investigations) | 1 | 0 | 0
Prostatic specific antigen increased (Investigations) | 0 | 0 | 1
Transaminases increased (Investigations) | 1 | 2 | 0
Varicella virus test positive (Investigations) | 0 | 0 | 1
Vitamin D decreased (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 5 | 4 | 4
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyper HDL cholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | 1 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Impaired fasting glucose (Metabolism and nutrition disorders) | 0 | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 2 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 8 | 9
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 4 | 6
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Chondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Enthesopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 4
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 10 | 2 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Torticollis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Elastofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Osteoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 4 | 3 | 5
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 1
Facial paralysis (Nervous system disorders) | 1 | 1 | 0
Headache (Nervous system disorders) | 15 | 12 | 17
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 4
Hypogeusia (Nervous system disorders) | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0
Meralgia paraesthetica (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 3 | 3 | 1
Motor dysfunction (Nervous system disorders) | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 1 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 0
Seizure like phenomena (Nervous system disorders) | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 1 | 1
Tension headache (Nervous system disorders) | 0 | 1 | 0
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 | 1 | 0
Affective disorder (Psychiatric disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 3 | 3 | 3
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1 | 0 | 1
Binge eating (Psychiatric disorders) | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 3 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 5 | 4
Mood altered (Psychiatric disorders) | 2 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1
Stress (Psychiatric disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Hypertonic bladder (Renal and urinary disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 0 | 2
Nocturia (Renal and urinary disorders) | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0
Polyuria (Renal and urinary disorders) | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 1
Renal cyst (Renal and urinary disorders) | 0 | 1 | 0
Urine odour abnormal (Renal and urinary disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 0 | 1
Breast cyst (Reproductive system and breast disorders) | 1 | 1 | 0
Breast disorder (Reproductive system and breast disorders) | 0 | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 3 | 0
Sexual dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 0 | 1
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 9
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 3
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 8
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 5 | 7
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Parapsoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 4
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 9 | 6 | 7
Rash (Skin and subcutaneous tissue disorders) | 4 | 0 | 5
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Trichorrhexis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Menopause (Social circumstances) | 0 | 0 | 1
Cataract operation (Surgical and medical procedures) | 0 | 0 | 1
Female sterilisation (Surgical and medical procedures) | 0 | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 11 | 7 | 7
Hypotension (Vascular disorders) | 0 | 1 | 0
Peripheral venous disease (Vascular disorders) | 0 | 0 | 1
Varicose vein (Vascular disorders) | 0 | 1 | 0
Vasodilatation (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2016-08-31): https://cdn.clinicaltrials.gov/large-docs/90/NCT02376790/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-06): https://cdn.clinicaltrials.gov/large-docs/90/NCT02376790/SAP_001.pdf